CLINICAL TRIAL: NCT04643093
Title: Orient Pharma Co., Ltd.
Brief Title: Compare the Efficacy and Safety of 1PC111 With Pitavastatin and Ezetimibe in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OP-1PC111-301
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemias
Keywords: Primary Hypercholesterolemia; Mixed Dyslipidemias
MeSH Terms: interventions — pitavastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pitavastatin (Active Comparator): Pitavastatin
  Interventions: Drug: Pitavastatin
- Ezetimibe (Active Comparator): Ezetimibe
  Interventions: Drug: Ezetimibe
- 1PC111 (Experimental): 1PC111
  Interventions: Drug: 1PC111

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin, QD
  Arms: Pitavastatin
Drug: Ezetimibe — Ezetimibe, QD
  Arms: Ezetimibe
Drug: 1PC111 — 1PC111, QD
  Arms: 1PC111

SUMMARY:
The study is to evaluate whether the efficacy of 1PC111 is superior to pitavastatin and ezetimibe in patients with primary hypercholesterolemia or mixed dyslipidemia in the 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hypercholesterolemia or mixed dyslipidemia
2. Subject meeting All of the following diagnoses at Baseline visit:

   * TG≦350 mg/dL
   * ALT and AST≦ 2.5 times of upper limit of normal (ULN) with no acute liver disease
   * Creatine kinase (CK) concentration≦2 times of UL N
   * Creatinine≦1.5 mg/dL
3. Subject who is willing and able to provide inform ed consent

Exclusion Criteria:

1. Female who is or intends to be pregnant or breast feeding, or has childbearing potential but without effective contraception.
2. Subject with documented HIV
3. Subject with uncontrolled hypothyroidism according to the investigator's judgment
4. Subject with unstable cardiovascular disease (CVD), including but not limited to congestive heart failure (CHF) defined as New York Heart Association class III or IV, unstable angina, unstable arrhythmia according to the investigator's judgment
5. Subject with unstable hepatic or biliary disorders, including but not limited to acute hepatitis, acute exacerbation of chronic hepatitis, liver cirrhosis, liver cancer, jaundice , and chronic hepatitis B or C under antiviral therapy
6. Subject with the following medical histories:

   * History of malignancy, exceptions made for the following malignancies: a)those determined to be cured or in remission for ≥ 5 years, b) curatively resected basal cell or squamous cell skin cancers, c) cervical cancer in situ, or resected colonic polyps
   * Acute coronary syndrome with or without cardiac catheterization within the past 9 months
   * Therapeutic cardiac catheterization (due to reasons other than acute coronary syndrome) within the past 6 months
7. Any unstable comorbidities or clinical conditions , including laboratory abnormalities which could lead to unacceptable risk to subject or confound data interpretation , per investigatiors judgment
8. Use any lipid lowering agent within 6 weeks prior to initiating the study treatment ( recheck this criterion at Day 1)
9. Use cyclosporine within 6 weeks prior to initiating the study treatment (recheck this criterion at Day 1)
10. Use any investigational product within 6 weeks prior to initiating the study treatment ( recheck this criterion at Day 1)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
The efficacy of 1PC111 is superior to pitavastatin and ezetimibe in patients | 12 week treatment period

SECONDARY OUTCOMES:
The efficacy and safety profile of 1PC111 , pitavastatin and ezetimibe during the treatment period and 2 week follow up period. | 12 week treatment period

CONTACTS AND LOCATIONS:
Locations (34):
- Australia (4):
  - Paratus Clinical Research Western Sydney, Blacktown
  - Northern Beaches Clinical Research, Brookvale
  - Emeritus Research, Camberwell
  - Paratus Clinical Research Central Coast, Kanwal
- New Zealand (7):
  - Southern Clinical Trials - Waitemata Ltd., Auckland
  - Southern Clinical Trials Totara, Auckland
  - Southern Clinical Trials Group Ltd, Christchurch
  - Lakeland Clinical Trials Waikato, Hamilton
  - Southern Clinical Trials Tasman, Nelson
  - Lakeland Clinical Trials Rotorua, Rotorua
  - Culloden Research Ltd., Tauranga
- Taiwan (23):
  - Changhua Christian Hospital, Changhua
  - Chiayi Christian Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital of the C.G.M.F., Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Tainan Municipal Hospital (Managed By Show Chwan Medical Care Corporation), Tainan
  - Cathay General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tamsui Mackay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation- LinKuo Branch, Taoyuan District

REFERENCES:
- [Derived] Chou MT, McGirr A, Jong GP, Chao TH, Lee IT, Huang CY, Chen CP, Hsieh CH, Lu CH, Sheu WH. Effect of 1PC111, a Fixed-dose Combination of Pitavastatin and Ezetimibe, Versus Pitavastatin or Ezetimibe Monotherapy on Lipid Profiles in Patients With Hypercholesterolemia or Mixed Dyslipidemia: A Randomized, Double-blind, Multicenter, Phase III Study. Clin Ther. 2022 Oct;44(10):1272-1281. doi: 10.1016/j.clinthera.2022.08.006. Epub 2022 Aug 25. PMID 36030106